CLINICAL TRIAL: NCT00868764
Title: An Investigation on the Effect of Age and BMI on the Pharmacokinetics of Transdermal Granisetron
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 392MD/40/C
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pharmacokinetics
Keywords: Effect of age; Effect of body fat; Granisetron; Pharmacokinetic profile; Sancuso® patch; Transdermal
MeSH Terms: interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sancuso® patch (Experimental): Subjects receiving 1 Sancuso® patch worn for 7 days
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — 3.1 mg/24 hours; transdermal. One patch applied to healthy intact skin on the upper outer arm and worn for 7 days
  Other Names: Sancuso® patch; Granisetron Transdermal System

SUMMARY:
This study aims to evaluate the effect of age and BMI on the pharmacokinetics and safety of Sancuso®.

DETAILED DESCRIPTION:
Sancuso® (granisetron transdermal system [TDS] or patch) was approved by the United States (US) Food and Drug Administration (FDA) in September 2008, indicated for the prevention of nausea and vomiting in patients receiving moderately and/or highly emetogenic chemotherapy regimens of up to 5 consecutive days' duration.

While in vivo pharmacokinetic studies with Sancuso® in healthy adults and in subjects receiving chemotherapy have been conducted, there are limited data from subjects who have altered skin integrity due to advanced age or poor nutritional status related to chronic illness. In addition, available data suggest that granisetron is delivered into subcutaneous fat and is released from that compartment over time. It is possible that individuals with varying nutritional status and resultant differences in subcutaneous fat would have differences in pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

-- Healthy male or female subjects:

Part I

* Aged ≥ 65 years at screening
* Control group: aged ≥ 18 to 45 years at screening

Part II -- Aged between 18 and 60 years, inclusive, at screening

Part I

-- BMI between 20.0 and 29.9 kg/m², inclusive

Part II

* Underweight (BMI < 18.5 kg/m²) or obese (BMI between 30.0 and 39.9 kg/m², inclusive)
* Control group: BMI between 20.0 and 24.9 kg/m², inclusive

Exclusion Criteria:

* Current or previous disease, disorder, allergy or condition that could affect study conduct or laboratory assessments, or that presents undue risk from study medication or procedures.
* Physical examination or screening investigation result that indicates subject is unfit for study.
* Scarring on upper arms.
* Positive virology, urine drugs of abuse or pregnancy test result (female subjects of childbearing potential only).
* Recent use of prescribed or over-the-counter medication.
* Received an investigational drug within 3 months (90 days) prior to patch application.
* Loss of ≥ 400 mL of blood (e.g. been a blood donor) within the previous 3 months.
* Average weekly alcohol consumption > 21 units (males) or 14 units (females), or habitually smokes ≥ 5 cigarettes or equivalent tobacco per day within the 6 months before patch application.
* Lactating female subjects and female subjects of childbearing potential not willing to use an acceptable form of contraception during and for 90 days after the study.
* Employee of the investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that investigator or study centre, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of the granisetron patch in elderly subjects (Part 1) and in underweight and obese subjects (Part 2) | 0 to 216 hours post-dose

SECONDARY OUTCOMES:
Safety and tolerability of the granisetron patch in elderly subjects (Part 1) and in underweight and obese subjects (Part 2) | Up to 23 days post-dose
Patch adhesion and residual granisetron after patch use in elderly subjects (Part 1) and in underweight and obese subjects (Part 2) | 0 to 168 hours post-dose
PK profile of the granisetron patch in elderly subjects vs younger subjects (Part 1) and PK profile of the granisetron patch in underweight and obese subjects vs in subjects whose body mass index (BMI) is within the normal range (Part 2) | 0 to 216 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Mair, Principal Investigator — Syneos Health
Locations (1):
- Charles River Clinical Services Edinburgh Ltd, Edinburgh, United Kingdom